CLINICAL TRIAL: NCT03345368
Title: Effect of Repetitive Transcranial Magnetic Stimulation in Combination With a Low-carbohydrate Diet in Patients With Obesity: a Randomized Controlled Study
Brief Title: Effect of rTMS in Combination With a Low-carbohydrate Diet in Patients With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Ajusco Medio (Other)
Responsible Party: Principal Investigator, Dra. Monica Ambriz Tututi, Especialista en área de Salud, Hospital General Ajusco Medio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211-010-01-17
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Obesity; Anxiety
Keywords: transcranial magnetic stimulation; obesity; diet
MeSH Terms: conditions — Obesity; Anxiety Disorders | interventions — Transcranial Magnetic Stimulation; Diet

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to one of two groups: the experimental group receiving rTMS and a placebo group receiving sham rTMS. Both groups will be on the low-carb diet.
Who Masked: Participant
Masking Description: Sham rTMS will be administered with the coil held in contact with the head but at 180 degrees from scalp to avoid stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS treated group (Experimental): A Magstim Rapid2 Stimulator equipped with a double 70mm alpha coil P/N 3191-00 (Magstim, Wales, UK) will be used to stimulate the motor cortex. Transcranial magnetic stimulation will be applied through a coil at 10 Hz, a field intensity of 90% of the motor threshold. Stimuli will be provided in 10 trains of 100 pulses, followed by a 28 s rest period.
  Interventions: Device: rTMS; Other: Diet
- sham rTMS group (Sham Comparator): Sham rTMS will be administered with the coil held in contact with the head but a 180 degrees from scalp, and the power parameter will be reduced by half to avoid stimulation.b
  Interventions: Device: sham rTMS; Other: Diet

INTERVENTIONS:
Device: rTMS — Patients will be stimulated in the dorso lateral frontal cortex. First, the motor threshold will be determined for each patient. To induce currents to the left primary sensory-motor cortex hand area (M1/S1) the coil will be placed over the scalp oriented at 45 ° from the mid-sagittal plane while subjects will sit comfortably on a chair. The coil will be systematically moved in this area until a contraction of the abductor will be identified. Motor evoked potentials (MEPs). MEPs will be registered with surface electrodes on the left hand abductor pollicis muscle using the same Magstim equipment. Then the parameters will be adjusted for the stimulation as was described before.
  Other Names: repetitive transcranial magnetic stimulation
  Arms: rTMS treated group
Device: sham rTMS — As well as the rTMS group, the motor threshold of each patient will be determined. They will experience a similar rTMS session with the difference that they not will be stimulated.
  Other Names: placebo
  Arms: sham rTMS group
Other: Diet — This intervention will be applied to both groups, rTMS and sham group, as a combined therapy. The diet is low in carbohydrates, like sugary foods, pasta and bread. Instead, patients eat food with protein, natural fats and vegetables.
  Other Names: conventional treatment

SUMMARY:
In the present study the investigators want to evaluate if the application of rTMS can reduce the anxiety and craving in patients with obesity helping them to follow a low carb-diet, as well as, to assess the changes in weight, body mass index and quality of life before and after rTMS or sham rTMS.

DETAILED DESCRIPTION:
Participants completed a written, informed consent and rTMS adult safety questionnaire. The inclusion criteria are:

individuals between 25 and 60 years of age with obesity in stage 1, 2 or 3. The exclusion criteria were: subjects with metabolic disorders, neurological condition, epilepsy, or pregnancy. The study conformed to the Declaration of Helsinki and was approved by the Institutional Medical Research Ethics Committee (Hospital Ajusco Medio, Mexico DF). The protocol will be applied as follows: 10 rTMS or sham sessions during two weeks. Following these two week, patients will receive 8 more sessions on weeks 4, 6, 8, 10, 12, 16, 20 and 24. Diet will be indicated during all the protocol. The sham group will receive sham rTMS sessions for two weeks, the additional sessions will be performed in the same manner thar in rTMS group.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30

Exclusion Criteria:

* Thyroid problems, anorexia, bulimia, epilepsy, schizophrenia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Obesity, changes in the body mass index | 7 days
  Obesity is a body mass index greater than or equal to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Ambriz-Tututi, Dr., Study Director — HospitalGeneral Ajusco Medio
Locations (1):
- Hospital General Ajusco Medio, México, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after study conclusion

REFERENCES:
- [Background] Alonso-Alonso M, Pascual-Leone A. The right brain hypothesis for obesity. JAMA. 2007 Apr 25;297(16):1819-22. doi: 10.1001/jama.297.16.1819. No abstract available. PMID 17456824
- [Background] Kober H, Mende-Siedlecki P, Kross EF, Weber J, Mischel W, Hart CL, Ochsner KN. Prefrontal-striatal pathway underlies cognitive regulation of craving. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14811-6. doi: 10.1073/pnas.1007779107. Epub 2010 Aug 2. PMID 20679212
- [Result] Barth KS, Rydin-Gray S, Kose S, Borckardt JJ, O'Neil PM, Shaw D, Madan A, Budak A, George MS. Food cravings and the effects of left prefrontal repetitive transcranial magnetic stimulation using an improved sham condition. Front Psychiatry. 2011 Mar 14;2:9. doi: 10.3389/fpsyt.2011.00009. eCollection 2011. PMID 21556279
- [Result] Uher R, Yoganathan D, Mogg A, Eranti SV, Treasure J, Campbell IC, McLoughlin DM, Schmidt U. Effect of left prefrontal repetitive transcranial magnetic stimulation on food craving. Biol Psychiatry. 2005 Nov 15;58(10):840-2. doi: 10.1016/j.biopsych.2005.05.043. Epub 2005 Aug 8. PMID 16084855